CLINICAL TRIAL: NCT04869631
Title: Screening for Amyloidosis Before Aortic Valve Elective Replacement (SAVER)
Brief Title: Screening for Amyloidosis Before Aortic Valve Elective Replacement
Acronym: SAVER
Status: Active, not recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Herzzentrum Berlin, Klinik für Innere Medizin - Kardiologie (Unknown); Klinik für Neurologie mit Experimenteller Neurologie, Charité - Universitätsmedizin Berlin (Unknown)
Responsible Party: Principal Investigator, Isabel Mattig, Project lead, Charite University, Berlin, Germany
Other Study IDs: EA4/235/20
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Amyloidosis; Aortic Valve Stenosis
Keywords: Cardiac Amyloidosis; Transthyretin Amyloidosis; ATTR; Aortic Stenosis; Screening
MeSH Terms: conditions — Amyloidosis; Aortic Valve Stenosis; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Aortic valve stenosis undergoing aortic valve replacement: Aortic valve stenosis undergoing aortic valve replacement.
  Interventions: Other: The outcome of an intervention is not evaluated, but aortic stenosis and additional amyloidosis are compared.

INTERVENTIONS:
Other: The outcome of an intervention is not evaluated, but aortic stenosis and additional amyloidosis are compared. — We aim to compare patients with aortic valve stenosis with and without cardiac amyloidosis.

SUMMARY:
Previous studies detected that up to 15% of patients undergoing aortic valve replacement (AVR) for degenerative aortic stenosis have concomitant transthyretin amyloidosis (ATTR) cardiomyopathy (Castano, 2017). The aim of this study is to investigate the effectivity and practicability of a systematic ATTR-Screening in patients undergoing planned AVR. Moreover, we plan to develop a screening algorithm to detect ATTR in aortic stenosis (AS).

DETAILED DESCRIPTION:
Untreated cardiac amyloidosis is accompanied with an impaired prognosis. Amyloidosis is often associated with ventricular hypertrophy which leads to severe heart failure and occurs frequently in conjunction with bradycardic or tachycardic malignant arrhythmia. Patients with degenerative aortic valve stenosis suffer more frequently from cardiac ATTR. However, it remains unclear whether the development of aortic stenosis is promoted by ATTR. Due to very similar symptoms (shortness of breath during physical exertion, reduced walking distance) diagnosis of aortic valve stenosis is more often diagnosed in a typical cohort of patients aged between 70-80 years but, in contrast, leads to underdiagnosis of patients with additional cardiac amyloidosis. Six to fifteen percent of patients with aortic valve replacement due to degenerative aortic valve stenosis exhibit a cardiac amyloidosis. Since cardiac amyloidosis without therapeutic intervention is associated with significantly reduced life expectancy, it can be assumed that these patients will not benefit to the same extent from the AVR alone as patients without ATTR. New therapeutic approaches for patients exhibiting ATTR lead to a reduction of mortality and hospitalizations. The primary aim of this study is to establish a simple ATTR screening tool in patients with planned AVR in the clinical routine and, furthermore, to compare the clinical course following AVR between patients with and without ATTR.

ELIGIBILITY:
Inclusion Criteria:

* age ≥40 years
* written informed consent from the patient or of his/her legal guardian
* hospitalization for AVR due to degenerative aortic valve stenosis

Exclusion Criteria:

* hemodynamically unstable patient
* severe co-morbidities with an estimated life expectancy of <1 year

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >40 years with aortic valve stenosis who are scheduled to undergo interventional or surgical aortic valve replacement at Deutsches Herzzentrum Berlin or Charité - Universitätsmedizin Berlin during a recruiting period of 18 months; in total approximately 1500 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number/ proportion of ATTR cases identified by systematic screening | Enrolment period: 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Kerr D. Lin zhong guan huai: terminal care in China. Am J Hosp Palliat Care. 1993 Jul-Aug;10(4):18-26. doi: 10.1177/104990919301000407. No abstract available. PMID 7687139
- [Background] Amramy A. Waste treatment for ground water recharge. Air Water Pollut. 1965 Oct;9(10):605-19. No abstract available. PMID 5837725
- See also: Amyloidosis center of the Charité — https://amyloidosis-center.charite.de/